CLINICAL TRIAL: NCT02771184
Title: Computerized Lung Sound Analysis
Acronym: CLSA
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Smolle-Juettner Freyja, Prof MD (Other)
Collaborators: Graz University of Technology (Other)
Responsible Party: Sponsor-Investigator, Smolle-Juettner Freyja, Prof MD, Univ.-Prof. Dr.med.univ., Medical University of Graz
Organization: Medical University of Graz (Other)
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Basic Science
Other Study IDs: 28-088 ex 15/16
Record Dates: First submitted 2016-04-22; First posted 2016-05-13 (Estimated); Last update posted 2019-05-20 (Actual); Status verified 2019-05

CONDITIONS: Pneumothorax; Pulmonary Fibrosis
MeSH Terms: conditions — Pneumothorax; Pulmonary Fibrosis

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (3):
- Lung-Healthy (Other): Subjects with no diagnosed lung disease. The intervention is the recording of lung sounds with the Lung Sound Recording System.
  Interventions: Device: Lung Sound Recording System
- Pneumothorax (Other): Subjects with pneumothorax. The intervention is the recording of lung sounds with the Lung Sound Recording System.
  Interventions: Device: Lung Sound Recording System
- Pulmonary Fibrosis (Other): Subjects with pulmonary fibrosis. The intervention is the recording of lung sounds with the Lung Sound Recording System.
  Interventions: Device: Lung Sound Recording System

INTERVENTIONS:
Device: Lung Sound Recording System — The lung sounds are recorded over the posterior chest in supine position on an examination table. A foam pad with several lung sound transducers is placed under the back of the subjects. During the recording the subjects wear a nose clip and hold a pneumotachograph with both hands. The subjects are instructed to breath at a certain airflow rate during inspiration, with natural breathing during expiration. Therefore, they receive a real-time feedback for the airflow rate. The airflow signal and the lung sounds from 16 lung sound transducers are recorded simultaneously for 30 seconds.

SUMMARY:
This clinical trial is conducted within the research project 'Computerized Lung Sound Analysis'. The research goal is the development of a system enabling the automatic classification of lung sounds, which will result in a decision support system for physicians.

The objective of this trial is to create a small lung sound corpus, enabling the development of a prototype of the described system. Therefore, investigators record lung sounds with several lung sound transducers distributed on the posterior chest of human test subjects.

DETAILED DESCRIPTION:
In this clinical trial investigators record lung sounds over the posterior chest of human test subjects. The subjects are either lung-healthy (control group) or subjects with pneumothorax condition or pulmonary fibrosis. The lung sounds are recorded in supine position on an examination table. A foam pad with several lung sound transducers is placed under the back of the subjects. During the recording the subjects wear a nose clip and hold a pneumotachograph with both hands. The subjects are instructed to breath at a certain airflow rate during inspiration, with natural breathing during expiration. For each subject investigators simultaneously record 30 seconds of the airflow signal and the lung sounds from 16 lung sound transducers.

ELIGIBILITY:
Inclusion Criteria:

General:

* Smoker and non-smoker
* 'Lung-healthy' subjects (control group), subjects with pneumothorax or subjects with pulmonary fibrosis

Additional for 'lung-healthy' subjects:

* COPD < 3 (GOLD Criteria)

Exclusion Criteria:

General:

* Body Mass Index > 30
* Preceding thoracic surgery
* Non-cooperation of the subject
* Intubated or tracheostomized subjects

Additional for 'lung-healthy' subjects:

* Disease of the respiratory system
* Taking medication influencing the respiration

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 24 (Actual)
Dates: Start 2016-04; Primary Completion 2018-03 (Actual); Study Completion 2018-03 (Actual)

PRIMARY OUTCOMES:
16-Channel Lung Sound Recordings and synchronous Airflow Recording | 30 Seconds
  The lung sounds and the airflow signal are simultaneously recorded with the Lung Sound Recording System. One time frame contains several breathing phases. Depending on the lung disease normal lung sounds are either altered or adventitious lung sounds are superimposed.

CONTACTS AND LOCATIONS:
Overall Officials: Freyja-Maria Smolle-Juettner, Univ.-Prof., Principal Investigator — Medical University of Graz
Locations (1):
- Medical University of Graz, Graz, Austria

IPD SHARING:
Plan to Share IPD: No